CLINICAL TRIAL: NCT04339530
Title: Association Between Vitamin D Status and Risk of Type 2 Diabetes in a Population of UK Adults: A Cross-sectional Study.
Brief Title: Vitamin D and Type 2 Diabetes Risk in UK Adults
Status: Suspended | Type: Observational
Why Stopped: This study is suspended until further notice. Recruitment should resume when COVID-19 safety restrictions are lifted.
Sponsor: Liverpool Hope University (Other)
Responsible Party: Principal Investigator, Grace Farhat, Principal Investigator, Liverpool Hope University
Other Study IDs: 7062019
Record Dates: First submitted 2020-04-03; First posted 2020-04-09 (Actual); Last update posted 2021-05-10 (Actual); Status verified 2021-05

CONDITIONS: Overweight; Obesity
Keywords: Vitamin D; Type 2 diabetes; Insulin resistance; Glucose
MeSH Terms: conditions — Overweight; Obesity; Diabetes Mellitus, Type 2; Insulin Resistance

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Normal weight and overweight adults — Association between vitamin D levels and insulin resistance

SUMMARY:
This study is exploring the association between vitamin D and Type 2 diabetes risk in normal weight and overweight UK adults.

DETAILED DESCRIPTION:
The aim of this study is to assess the link between vitamin D status and glucose homeostasis in a population of normal weight and overweight individuals (BMI> 18.5 Kg/m2).

ELIGIBILITY:
Inclusion Criteria:

* Normal weight and overweight and obese adults (BMI>= 18.5 Kg/m2) with no restriction to ethnicity, occupation or socioeconomic status.
* Males and females
* 18-50 years

Exclusion Criteria:

* Patients diagnosed with diabetes type 2, myocardial infarction or coronary heart disease.
* HbA1c > 6.4%
* Pregnancy
* Diagnosis of liver disease (including liver enzymes > 3 times above normal values)
* Diagnosis of renal disease (creatinine of > 150 mmol/l)
* Post-menopausal women

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Overweight and obese adults , aged 18-50 (premenopausal women), males and females with no known chronic conditions.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2022-07-01 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
HOMA-IR (Homeostasis modelling assessment-Insulin resistance) | One venous sample collected after 8 hours of fasting
  A venous blood sample collected for the measurement of insulin and glucose levels.

SECONDARY OUTCOMES:
Fasting bood glucose levels | One venous sample collected after 8 hours of fasting
  A venous blood sample collected for the measurement of glucose levels
HbA1C | Sample collected at one single time point with no follow-up
  Fingerprick sample
Body fat percentage | Measurement conducted in the morning after 8 hours of fasting
  Body fat percentage measured through DEXA
Central and brachial Systolic and Diastolic Blood pressure | Measurement taken 3 times after a-10 minute rest
  Blood pressure measured using a digital sphygmomanometer
Augmentation index | Measurement taken 3 times after a-10 minute rest
  Arterial stiffness assessment test

CONTACTS AND LOCATIONS:
Locations (1):
- School of Health sciences, Liverpool, United Kingdom

IPD SHARING:
Plan to Share IPD: No